CLINICAL TRIAL: NCT00265785
Title: Phase II Trial of Pemetrexed in Patients With Selected Stage IIIB and IV Bronchioloalveolar Carcinoma (BAC)
Brief Title: S0526: Pemetrexed Disodium in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to poor accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000456424; U10CA032102 (NIH); S0526 (Other: SWOG)
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Results first posted 2012-11-01 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Lung Cancer
Keywords: bronchoalveolar cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed (Experimental): pemetrexed
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — Pemetrexed 500 mg/m^2 intravenous (IV) over 10 min every 21 days until any of the following criteria is met: (1) Progression of disease or symptomatic deterioration; (2) Unacceptable toxicity; (3) Treatment delay ≥ 3 weeks, for any reason; (4) The patient may withdraw from the study at any time for any reason; (5) Physician's discretion.
  Other Names: Alimta

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pemetrexed disodium, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pemetrexed disodium may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well pemetrexed disodium works in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess overall survival of patients with selected stage IIIB or IV bronchoalveolar carcinoma treated with pemetrexed disodium.

Secondary

* Evaluate the progression-free survival of patients treated with this drug.
* Evaluate the response rate (confirmed and unconfirmed, partial and complete) in the subset of patients with measurable disease treated with this drug using standard RECIST criteria and computer assisted image analysis.
* Evaluate frequency and severity of toxicities in patients treated with this drug.
* Perform molecular correlative studies on patient tissue to investigate potential predictors of efficacy. (This will not be completed as this study was closed due to poor accrual.)

OUTLINE: Patients are stratified according to prior treatment with gefitinib or erlotinib (yes vs no).

Patients receive pemetrexed disodium intravenous (IV) on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 3 years.

PROJECTED ACCRUAL: A total of 99 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed bronchoalveolar carcinoma (BAC) or BAC variants such as adenocarcinoma with BAC features or BAC with invasive adenocarcinoma

  * Cytology specimens, such as bronchial brushings, washings, or fine needle aspiration specimens alone are not acceptable for diagnosis
* Stage IV disease OR selected stage IIIB (T4 [secondary to malignant pleural effusion only], any N, M0) disease
* Incompletely resected or unresectable disease
* Pleural effusions, ascites, or laboratory parameters cannot be only evidence of disease
* Measurable disease or nonmeasurable disease documented by CT scan
* No known brain metastases

PATIENT CHARACTERISTICS:

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT and SGPT ≤ 2.5 times ULN ( ≤ 5 times ULN if due to liver metastases)
* Alkaline phosphatase ≤ 2.5 times ULN ( ≤ 5 times ULN if due to bone metastases)
* Creatinine clearance ≥ 45 mL/min OR creatinine ≤ 1.5 times ULN
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm³
* Zubrod 0-2
* No history of allergic reaction to compounds of similar chemical or biological composition as pemetrexed disodium
* Must provide smoking history
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Able to swallow pills

PRIOR CONCURRENT THERAPY:

* No more than 2 prior systemic therapies (including epidermal growth factor receptor inhibitor)
* At least 28 days since prior systemic therapy
* Patients treated with prior erlotinib or gefitinib must have shown progression since treatment
* No prior pemetrexed disodium
* At least 28 days since prior radiotherapy and recovered

  * Must have measurable or nonmeasurable disease outside previously irradiated area or a new lesion within previously irradiated area
* At least 14 days since prior palliative radiotherapy and recovered
* At least 28 days since prior thoracic or major surgery and recovered
* No concurrent surgery
* No other concurrent therapy (hormonal, biologic or radiotherapy) for this disease
* No concurrent antiretroviral therapy
* Patients should discontinue non-steroidal anti-inflammatory drugs (NSAIDs) with longer half lives (etodolac, ketordac, sulindac, naproxen, naproxen sodium, oxaprozin, nabumetone, diflunisal, salsalate, celecoxib, rofecoxib, valdecoxib, meloxicam, piroxicam) at least 5 days before and for 2 days following pemetrexed treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derick H. Lau, MD, Principal Investigator — University of California, Davis; Rachel E. Sanborn, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (112):
- United States (112):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - NEA Medical Center - Stadium Boulevard, Jonesboro, Arkansas
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Cancer Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Danville Regional Medical Center, Danville, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed: Pemetrexed Disodium 500 mg/m^2 intravenous (IV) over 10 min every 21 days until any of the following criteria is met: (1) Progression of disease or symptomatic deterioration; (2) Unacceptable toxicity; (3) Treatment delay ≥ 3 weeks, for any reason; (4) The patient may withdraw from the study at any time for any reason; (5) Physician's discretion.
Period: Overall Study
Arm/Group | Pemetrexed
Started | 27
Eligible | 26
Eligible and Began Protocol Treatment | 24
Completed | 0
Not Completed | 27
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 3
Not completed — Progression/Relapse | 15
Not completed — Not protocol specified | 2
Not completed — Ineligible | 1
Not completed — Did not receive protocol treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 24
Age Continuous [Median (Full Range); unit: years] | 68.2 [49.6 to 82.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 1
  Unknown or Not Reported | 1
Histology [Number; unit: participants]
  Adenocarcinoma w/BAC features | 18
  Bronchioloalveolar | 6
Number of Metastatic Sites [Number; unit: participants]
  Single | 12
  Multiple | 7
  None | 5
Stage [Number; unit: participants]
  IIIB | 0
  IV | 24
Prior EGFR-TKI Therapy [Number; unit: participants]
  No | 19
  Yes | 5
Prior Radiation Therapy [Number; unit: participants]
  Yes | 3
  No | 21
Prior Systemic Treatment [Number; unit: participants]
  Yes | 10
  No | 14
Prior Surgery [Number; unit: participants]
  Yes | 11
  No | 13
Zubbrod Performance Status [Number; unit: participants] — Performance status is graded according to the Zubrod Performance Status Scale. Patients with a performance status of 0 are fully active, able to carry on all pre-disease performance without restriction. Patients with a performance status of 1 are restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  participants
    0 | 12
    1 | 12
Smoking Status [Number; unit: participants]
  Current | 5
  Former | 16
  Never | 3
Weight Loss Last 6 months [Number; unit: participants]
  < 5% | 20
  5% to < 10% | 3
  10% to 20% | 1
  > 20% | 0

OUTCOME MEASURES:

1. Secondary Outcome: Progression-free Survival
Description: Progression is defined as any one or more of the following: 20% increase in the sum of longest diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline; Unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided); Appearance of any new lesion/site; Death due to disease without prior documentation of progression and without symptomatic deterioration. Symptomatic deterioration is defined as globabl deterioration of health status requiring discontinuation of treatment without objective evidence of progression. Progression-free survival is measured from date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression-free are censored at date of last contact.
Time Frame: 0 - 3 years
Population: Eligible and analyzable patients were included in this measure.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Premetrexed: Pemetrexed Disodium 500 mg/m^2 intravenous (IV) over 10 min every 21 days until any of the following criteria is met: (1) Progression of disease or symptomatic deterioration; (2) Unacceptable toxicity; (3) Treatment delay ≥ 3 weeks, for any reason; (4) The patient may withdraw from the study at any time for any reason; (5) Physician's discretion.
Arm/Group | Premetrexed
Number analyzed (Participants) | 24
months | 6 [3 to 14]

2. Primary Outcome: Overall Survival
Description: Measured from date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: 0 - 3 years
Population: Eligible and analyzable patients were included in this measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Premetrexed
Number analyzed (Participants) | 24
months | 25 [15 to 36]

3. Secondary Outcome: Response (Confirmed and Unconfirmed, Complete and Partial)
Description: Complete response (CR) is complete disappearance of all measurable and non-measurable disease. No new lesions. No disease related symptoms. Normalization of markers and other abnormal lab values. Partial Response (PR) is greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. Confirmation of CR or PR means a repeat scan at least 4 weeks apart documented before progression or symptomatic deterioration.
Time Frame: Assessed at weeks 7 and 13 while on treatment. After off treatment prior to disease progression, disease assessment takes place every 3 months for a maximum of 3 years.
Population: Eligible and analyzable patients with measurable disease at baseline are included in this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Premetrexed
Number analyzed (Participants) | 17
percentage of participants | 29 [10 to 56]

4. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 3.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Patients were assessed for adverse events 4 weeks after starting treatment. Assessments for adverse events continued after every cycle of treatment (every 3 weeks) for the duration of protocol treatment.
Population: Eligible patients who received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Premetrexed
Number analyzed (Participants) | 24
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 1
  AST, SGOT | 1
  Diarrhea | 1
  Dyspnea (shortness of breath) | 1
  Fatigue (asthenia, lethargy, malaise) | 3
  Febrile neutropenia | 1
  Glucose, serum-high (hyperglycemia) | 3
  Hemoglobin | 2
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Bronchus | 1
  Leukocytes (total WBC) | 2
  Lymphopenia | 1
  Neutrophils/granulocytes (ANC/AGC) | 3
  Platelets | 2

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events after completion of each cycle of treatment.
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 22/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed (N=24)
Hemoglobin (Blood and lymphatic system disorders) | 13
Constipation (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 7
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 2
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 6
Edema: limb (General disorders) | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 16
Fever (in the absence of neutropenia, where neutropenia is defined as ANC lt1.0 x 10e9/L) (General disorders) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 13
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 9
Alkaline phosphatase (Investigations) | 5
Leukocytes (total WBC) (Investigations) | 3
Lymphopenia (Investigations) | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 5
Platelets (Investigations) | 3
Weight gain (Investigations) | 2
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 8
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 7
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3
Neuropathy: sensory (Nervous system disorders) | 2
Pain - Head/headache (Nervous system disorders) | 5
Taste alteration (dysgeusia) (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 4
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No